CLINICAL TRIAL: NCT03702205
Title: The Effect of Betaine Supplementation on Body Composition and Physical Capacity of Speed-strength Male Athletes
Brief Title: Betaine Effect in Speed-strength Athletes
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Life Sciences (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ULS00005
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Supplementation; Sport

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Betaine supplementation (Experimental): The experimental procedure for each athlete includes a 3-week betaine supplementation either 2.5 g or 5 g daily. Betaine will be administered in the form of capsules containing either 0.5 or 1 g betaine. The capsules will be ingested with at least 250 mL of water. Each athlete will ingest 5 betaine capsules a day. On training days the supplements will be taken in the morning (2 capsules), in the evening (2 capsules) and 1.5 hours before training session (1 capsule). On rest days the supplements will be taken in the morning (2 capsules), in the afternoon (1 capsule) and in the evening (2 capsules).
  Interventions: Dietary Supplement: Betaine supplementation; Dietary Supplement: Placebo treatment
- Placebo treatment (Experimental): The experimental procedure for each athlete included a 3-week placebo administration. Placebo will be capsules with starch. Placebo will be ingested with at least 250 mL of water. Each athlete will ingest 5 placebo capsules a day. On training days the supplements will be taken in the morning (2 capsules), in the evening (2 capsules) and 1.5 hours before training session (1 capsule). On rest days the supplements will be taken in the morning (2 capsules), in the afternoon (1 capsule) and in the evening (2 capsules).
  Interventions: Dietary Supplement: Betaine supplementation; Dietary Supplement: Placebo treatment

INTERVENTIONS:
Dietary Supplement: Betaine supplementation — Group taking oral betaine supplementation
Dietary Supplement: Placebo treatment — Group taking oral supplementation with placebo (starch) in a similar capsule form.

SUMMARY:
The study is aimed at assessing the influence of two betaine doses (2.5 g∙d-1 and 5 g∙d-1) supplemented for three weeks in a group of speed-strength trained athletes on anaerobic capacity in Wingate test, performance in CrossFit-like exercise test - Fight Gone Bad, alterations in body compositions and total body water.

DETAILED DESCRIPTION:
The main aim of the project is the assessment of the effects of 3 weeks supplementation with two doses of betaine (2.5 g∙d-1 and 5 g∙d-1) on anaerobic capacity, CrossFit performance, body composition, and betaine metabolism in a group of male speed-strength trained athletes.

The study is designed as a double-blind, randomized, placebo-controlled crossover trial. 80 male participants will be divided randomly into two parallel groups: one receiving 2.5 g·d-1 betaine and the second receiving 5 g·d-1 betaine. In both experimental groups participants will receive both betaine supplement or placebo in a random order. The supplementation periods (betaine and placebo) will last for three weeks each and will be separated by a 3-week washout. The participants will attend four study meetings at the Institute of Human Nutrition and Dietetics, Poznan University of Life Sciences, Poland. Food intake before and during the intervention will be assessed with the use of food diary and intakes of macro- and micronutrients will be calculated with the use of Dieta 5.0 software. On each visit Wingate ergocycling test will be performed, body composition will be measured and blood samples will be taken. The same day in the afternoon/evening hours the Fight Gone Bad (FGB) test will be performed. Body composition will be assessed based on air displacement plethysmography technology using the Bod Pod®. Moreover, total body water content will be analyzed by bioelectric impedance with the use of a BIA 101S analyzer. Anaerobic capacity will be assessed using the classical Wingate test on a cycloergometer. In order to assess CrossFit performance the FGB test will be performed. In blood samples the investigators plan to analyze concentrations of: lipoproteins and triglycerides (biochemical analyzer), betaine (LC-MS method), amino acid profile (LC-MS method), and testosterone (ELISA). MTHFR genotype will be analyzed with using a PCR-RFLP method. Data will be analyzed using the STATISTICA 12 software program.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from all participants before the study
* a current medical clearance to practice sports,
* training experience: at least 1 year (of CrossFit ttraining),
* minimum of 2 workout sessions (combat sport) a week,

Exclusion Criteria:

* current injury,
* any health-related contraindication,
* declared general feeling of being unwell,
* unwilling to follow the study protocol,
* serious disease or metabolic problems,
* intake of betaine, choline or creatine supplements 4 weeks before the beginning of the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-06-20 (Estimated); Study Completion 2021-10-12 (Estimated)

PRIMARY OUTCOMES:
Changes in fat mass and fat free mass after betaine supplementation | Baseline and after 3 weeks
  Fat mass (kg) and fat free mass (kg) analysis
Changes in anaerobic capacity after betaine supplementation | Baseline and after 3 weeks
  The Wingate cycling test (W)
Changes in specific performance capacity after betaine supplementation | Baseline and after 3 weeks
  The CrossFit-specific physical fitness test: Fight Gone Bad (reps.)

SECONDARY OUTCOMES:
Changes in total body water after betaine supplementation | Baseline and after 3 weeks
  Total body water content (%)
Changes in testosterone level (ng/L) after betaine supplementation | Baseline and after 3 weeks
  Testosterone level (ng/L)
Changes in amino acid profile after betaine supplementation | Baseline and after 3 weeks
  Amino acid profile (μmol/L)
Changes in blood betaine | Baseline and after 3 weeks
  Blood betaine (µmol/L)
Changes in total, LDL and HDL cholesterol and triacylglycerol after betaine supplementation | Baseline and after 3 weeks
  Total, LDL and HDL cholesterol (mg/dL) and triacylglycerol (mg/dL)
Difference in response to betaine supplementation depending on MTHFR (rs1801133) polymorphism | Baseline and after 3 weeks
  MTHFR (rs1801133) polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Agata Chmurzyńska, Professor, Study Director — Institute of Human Nutrition and Dietetics, Poznan University of Life Sciences, Poznan, Poland
Locations (1):
- Institute of Human Nutrition and Dietetics, Poznan University of Life Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zawieja E, Durkalec-Michalski K, Sadowski M, Glowka N, Chmurzynska A. Betaine supplementation improves CrossFit performance and increases testosterone levels, but has no influence on Wingate power: randomized crossover trial. J Int Soc Sports Nutr. 2023 Dec;20(1):2231411. doi: 10.1080/15502783.2023.2231411. PMID 37409757